CLINICAL TRIAL: NCT01917578
Title: Phase III Trail of Breast Cancer Shrinkage Modes After Neoadjuvant Chemotherapy With Whole-mount Serial Sections and Three-dimensional Pathological and MRI Reconstruction
Brief Title: Study of Breast Cancer Shrinkage Modes After Neoadjuvant Chemotherapy With Whole-mount Serial Sections and Three-dimensional Pathological and MRI Reconstruction
Acronym: BCSMANC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director, Head of Breast Cancer Center, Principal Investigator, Clinical Professor, Shandong Cancer Hospital and Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BCSMANC001
Record Dates: First submitted 2013-08-04; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; shrinkage modes; three-dimensional reconstruction; neoadjuvant chemotherapy; Magnetic Resonance Imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography; Biopsy, Large-Core Needle; Mastectomy, Segmental; Mastectomy, Modified Radical; Mammography; AC protocol; Cyclophosphamide; Doxorubicin; EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Half Cycles Group (Experimental): Patients complete half of the whole cycles of neoadjuvant chemotherapy.
  Interventions: Device: Ultrasound; Procedure: CNB; Procedure: BCS, Modified Radical Mastectomy; Device: Pathologic Large Tissue Selected Table; Device: Leica TP1020; Device: Pathologic Large Tissue Embedded Table; Device: Leica SM2000 R; Procedure: HE Stain; Device: CX22; Device: Epson V600; Procedure: Three-Dimensional Reconstruction; Device: Mammography; Drug: TAC,TC,TA,CAF,CEF
- Whole Cycles Group (Experimental): Patients complete whole cycles of neoadjuvant chemotherapy.
  Interventions: Device: Ultrasound; Procedure: CNB; Procedure: BCS, Modified Radical Mastectomy; Device: Pathologic Large Tissue Selected Table; Device: Leica TP1020; Device: Pathologic Large Tissue Embedded Table; Device: Leica SM2000 R; Procedure: HE Stain; Device: CX22; Device: Epson V600; Device: MRI; Procedure: Three-Dimensional Reconstruction; Device: Mammography; Drug: AC-P,TEC,AC,TC,TCH,CEF,TAC,CAF

INTERVENTIONS:
Device: Ultrasound — 1. Evaluation of the tumor size by sonography is performed before neoadjuvant chemotherapy and prior to surgery.
  2. Measurement of tumor size refers to WHO standards.
  Other Names: GE LOGIQ C5
Procedure: CNB — Typically, the pretreatment tumor specimen will be a core needle biopsy. Because 15% to 28% of patients will have no residual tumor after NAT, it is important to have an adequate pretreatment sample in which an unequivocal diagnosis of invasive carcinoma is established and evaluation of hormone receptors and HER2/ neu status is completed before treatment.
  Other Names: core needle biopsy
Procedure: BCS, Modified Radical Mastectomy — All patients after neoadjuvant chemotherapy are performed BCS and modified radical mastectomy.
  Other Names: BCS: breast conservative surgery
Device: Pathologic Large Tissue Selected Table — 1. Pathologic large tissue selected table has obtained Chinese patent.Its license ID is CN101261200.
  2. Each piece of breast tissues by cutting with the table has 3mm thickness.
Device: Leica TP1020 — Procedure:
  1. Alcohol 70 % 1h
  2. Alcohol 80 % 1h
  3. Alcohol 85 % 1h
  4. Alcohol 90 % 1h
  5. Alcohol 95 % 1h
  6. Alcohol Ⅰ 100 % 1h
  7. Alcohol Ⅱ 100 % 1h
  8. Xylene Ⅰ 2h
  9. Xylene Ⅱ 2h
  10. Xylene Ⅲ 2h
  11. Paraffin 6h
  12. Paraffin 6h
  Other Names: Semi-enclosed Benchtop Tissue Processor Leica TP1020
Device: Pathologic Large Tissue Embedded Table — 1. The table is made of brass .It is applying for a chinese patent.
  2. The table can simultaneously embed 8 piece of breast tissues.
Device: Leica SM2000 R — Each of paraffin section has 4 um thickness.
  Other Names: Sliding microtome Leica SM2000 R
Procedure: HE Stain — Procedure:
  1. Xylene Ⅰ 60℃ 15-20 minutes
  2. Xylene Ⅱ 60℃ 15-20 minutes
  3. Alcohol 100% Ⅰ 3-5 minutes
  4. Alcohol 100% Ⅱ 3-5 minutes
  5. Alcohol 95% Ⅱ 3-5 minutes
  6. Alcohol 90% Ⅱ 3-5 minutes
  7. Wash in running tap water for 3 minutes
  8. Hematoxylin 5-10 minutes
  9. Wash in running tap water for 3 minutes
  10. Differentiate in 1% acid alcohol for 30 seconds
  11. Wash in running tap water for 1 minute
  12. Bluing in 0.2% ammonia water for 30-60 seconds
  13. Wash in running tap water for 3 minutes
  14. Counterstain in eosin Y solution for 30-60 seconds
  15. Wash in running tap water for 1 minute
  16. Alcohol 90% Ⅱ 2-3 minutes
  17. Alcohol 95% Ⅱ 2-3 minutes
  18. Alcohol 100% Ⅱ 3-5 minutes
  19. Alcohol 100% Ⅱ 3-5 minutes
  20. Xylene Ⅲ 5-10 minutes
  21. Xylene Ⅳ 5-10 minutes
  22. Mounting with neutral resin
Device: CX22 — The residual tumor areas are microscopically outlined on each slice by pathologist.
  Other Names: Biological Microscope CX22（Olympus）
Device: Epson V600 — 1. Each slice that has been microscopically outlined is scanned by Epson V600.
  2. Every image by scanning should be saved as JPG.
  Other Names: Epson Perfection V600 Photo Scanner
Device: MRI — 1. Evaluation of the tumor size by MRI was performed before neoadjuvant chemotherapy and prior to surgery.
  2. Measurement of tumor size refers to WHO standards.
  3. The images of patients which were scanned by MRI should be burned onto disc for 3d reconstruction.
  Other Names: Philips Achieva 3.0T MRI System
  Arms: Whole Cycles Group
Procedure: Three-Dimensional Reconstruction — A.Pathological images three-dimensional reconstruction:
  1. Pathological images registration is based on skin and shear mark by Photoshop 13.0 software.
  2. Residual tumor boundary on Pathological images after registration are outlined and taken three-dimensional reconstruction by 3D-doctor 4.0 software.
  3. Observe the shrinkage modes in three-dimensional space.
  4. According to WHO standard,the boundaries of all residual tumor images are displayed in one plane and the longest diameter and its longest perpendicular diameter of boundaries are measured in one-dimensional space.
  5. According to RECIST standard,the longest diameter of boundaries of residual tumor images in three-dimensional space.
  B.MRI images three-dimensional reconstruction:the procedure is similar to Pathological images three-dimensional reconstruction
Device: Mammography — 1. Evaluation of the tumor size by mammography is performed before neoadjuvant chemotherapy and prior to surgery.
  2. Measurement of tumor size and calcification extent refers to WHO standards.
  3. Calcification extent is not only measured in mammography image but also under microscope.
  Other Names: GE Mammography
Drug: TAC,TC,TA,CAF,CEF — 1. TAC:Docetaxel 75 mg/㎡ iv day 1 + Doxorubicin 50 mg/㎡ in day 1 + Cyclophosphamide 500 mg/㎡ iv day 1(Cycled every 21 days for 3 cycles)
  2. TC:Docetaxel 75 mg/㎡ iv day 1 + Cyclophosphamide 600 mg/㎡in day 1(Cycled every 21 days for 2 cycles)
  3. TA:Docetaxel 75 mg/㎡ iv day 1 + Doxorubicin 50 mg/㎡ in day 1(Cycled every 21 days for 2 cycles)
  4. CAF:Cyclophosphamide 100 mg/㎡ po days 1-14 + Doxorubicin 30 mg/㎡ iv days 1,8 +5-fluorouracil 500 mg/㎡ iv days 1,8(cycled every 28 days for 3 cycles)
  5. CEF:Cyclophosphamide 75 mg/㎡ po day 1-14 + Epirubicin 60 mg/㎡ iv days 1,8 + 5-fluorouracil 500mg/㎡ iv days 1,8(cycled every 28 days for 3 cycles)
  Other Names: 1.TAC(docetaxel/doxorubicin/cyclophosphamide); 2.TC(docetaxel/cyclophosphamide); 3.TA(paclitaxel/doxorubicin); 4.CAF(fluorouracil/doxorubicin/cyclophosphamide); 5.CEF(cyclophosphamide/epirubicin//fluorouracil)
  Arms: Half Cycles Group
Drug: AC-P,TEC,AC,TC,TCH,CEF,TAC,CAF — 1. AC-P:Doxorubicin 60 mg/㎡ iv day 1 +Cyclophosphamide 600 mg/㎡ iv day 1(Cycled every 14 days for 4 cycles)→ Paclitaxel 175mg/㎡ by 3h iv infusion day 1(Cycled every 14 days for 4 cycles) or Paclitaxel 80mg/㎡ by 1h iv infusion weekly for 12 wks.
  2. TEC:Docetaxel 75 mg/㎡ iv day 1 + Epirubicin 75 mg/㎡ in day 1 + Cyclophosphamide 500 mg/㎡ iv day 1(Cycled every 21 days for 6 cycles)
  3. AC:Doxorubicin 60 mg/㎡ in day 1 + Cyclophosphamide 600 mg/㎡ iv day 1(Cycled every 21 days for 4 cycles)
  4. TC:Docetaxel 75 mg/㎡ iv day 1 + Cyclophosphamide 600 mg/㎡in day 1(Cycled every 21 days for 4 cycles)
  5. TCH:Docetaxel 75 mg/㎡ iv day 1 + Carboplatin AUC 6 iv day1(Cycled every 21 days for 6 cycles) + Trastuzumab 4 mg/kg iv wk 1 → Trastuzumab 2 mg/kg iv for 17 wks → Trastuzumab 6 mg/kg iv every 3 wks to complete 1 year.
  6. CEF:Cyclophosphamide 75 mg/㎡ po day 1-14 + Epirubicin 60 mg/㎡ iv days 1,8 + 5-fluorouracil 500mg/㎡ iv days 1,8(cycled every 28 days for 6 cycles)
  Other Names: 1.AC(doxorubicin/cyclophosphamide)-P(paclitaxel); 2.TEC(docetaxel/epirubicin/cyclophosphamide); 3.AC(doxorubicin/cyclophosphamide)-T(docetaxel); 4.TC(docetaxel/cyclophosphamide); 5.TCH(docetaxel/carboplatin/trastuzumab); 6.CEF(cyclophosphamide/epirubicin/fluorouracil); 7.TAC(docetaxel/doxorubicin/cyclophosphamide); 8.CAF(fluorouracil/doxorubicin/cyclophosphamide)
  Arms: Whole Cycles Group

SUMMARY:
The main clinical goal of NAC is to down-stage the primary tumor for BCS,yet BCS after NAC has been associated with significantly higher ipsilateral breast tumor recurrences.The accuracy of breast tumor excision in BCS can dramatically reduce IBTR.The main reseason of IBTR might be the uncertain shrinkage modes of the breast cancer after NAC.This clinical trial is firstly carried out to make clear the shrinkage modes of the primary tumor after 3 cycles and whole cycles of NAC,respectively,with whole-mount serial section(WMSS) and three-dimensional(3D) pathological reconstruction of the residual tumor.The second objective is to investigate the predictive value of 3D MRI reconstruction for the shrinkage modes of the primary tumor after NAC.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients,locally advanced breast cancer,age ≥18 years.
2. Histologically confirmed invasive adenocarcinoma of the breast.
3. Primary palpable disease confined to a breast and axilla on physical examination. For patients without clinically suspicious axillary adenopathy, the primary tumor must be larger than 2 cm in diameter by physical exam or imaging studies (clinical T2-T3, N0-N1, M0). For patients with clinically suspicious axillary adenopathy, the primary breast tumor can be any size (clinical T1-3, N1-2, M0). (T1N0M0 lesions are excluded.)
4. Patients without clearly defined palpable breast mass or axillary lymph nodes but radiographically measurable tumor masses are acceptable. Accepted procedures for measuring breast disease are mammography, MRI, and breast ultrasound. This will need to be re-evaluated after 3 cycles and prior to surgery.
5. ECOG 0 or 2
6. No distant metastasis, as documented by complete staging workup ≤6 weeks prior to initiation of study treatment.
7. No previous treatment for breast cancer.
8. Adequate hematologic function with:

   Absolute neutrophil count (ANC) >1500/μL. Platelets ≥100,000/μL. Hemoglobin ≥10 g/dL.
9. Adequate hepatic function with:

   Serum bilirubin ≤ the institutional upper limit of normal (ULN). Aspartate aminotransferase (AST) ≤2.5 x institutional ULN. Alanine aminotransferase (ALT) ≤2.5 x institutional ULN.
10. Adequate renal function with serum creatinine ≤1.5 x ULN.
11. Planned primary systemic (neoadjuvant) chemotherapy and surgical resection of residual primary tumor (mastectomy or lumpectomy/breast conservation) following completion of neoadjuvant chemotherapy

Exclusion Criteria:

1. inflammatory breast cancer
2. Pregnancy or breast-feeding.A negative serum pregnancy test within 7 days prior to first study treatment (Day 1, Cycle 1) for all women of childbearing potential is required. Patients of childbearing potential must agree to use a birth control method that is approved by their study physician while receiving study treatment and for 3 weeks after their last dose of study treatment. Patients must agree to not breast-feed while receiving study treatment.
3. Concurrent treatment with an ovarian hormonal replacement therapy or with hormonal agents such as raloxifene, tamoxifen or other selective estrogen receptor modulator (SERM). Patients must have discontinued use of such agents prior to beginning study treatment.
4. Uncontrolled intercurrent illness including (but not limited to) ongoing or active infection.
5. Concurrent treatment with any anti-cancer therapy other than those agents used in this study.
6. Mental condition or psychiatric disorder that would prevent patient comprehension of the nature, scope, and possible consequences of the study or that would limit compliance with study requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2008-08; Primary Completion 2014-03 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
The shrinkage modes of breast tumor after NAC. | 6 year
  The tumor shrinkage modes of the primary tumor in patients with locally advanced breast cancer after 3 cycles and whole cycles of neoadjuvant chemotherapy(NAC).

SECONDARY OUTCOMES:
The WMSS and 3D pathological reconstruction of the residual tumors after NAC. | 6 year
  The whole-mount serial section(WMSS) and three-dimensional(3D) pathological reconstruction of the residual tumors after NAC.

OTHER OUTCOMES:
The predictive value of 3D MRI reconstruction for the shrinkage modes of primary tumor after NAC. | 4 year
  The predictive value of 3D MRI reconstruction for the shrinkage modes of the primary tumor after whole cycles of NAC.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-sheng Wang, MD, Study Chair — Shandong Cancer Hospital and Institute; Tao Yang, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China

REFERENCES:
- [Result] Y-S Wang, Z-P Zhang, G Liu, D-B Mu, and X-Y Sun.Study of Breast Cancer Shrinkage Modes After Neoadjuvant Chemotherapy With Whole-mount Serial Sections and Three-dimensional Pathological and MRI Reconstruction. Cancer Res 2012;72(24 Suppl):Abstract nr P1-14-17.